CLINICAL TRIAL: NCT07199725
Title: Clinical and Radiographic Evaluation of Natural Bovine Bone With Hyaluronic Acid on Osseointegration of Immediate Implant: A Randomized Clinical Study
Brief Title: Clinical and Radiographic Evaluation of Natural Bovine Bone With Hyaluronic Acid on Osseointegration of Immediate Implant.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, mohamed wageh foad, principal investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 544/2022
Record Dates: First submitted 2025-09-02; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Dental Implants
Keywords: immediate dental implants; natural bovine bone
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: This clinical study was conducted on 16 badly decayed single rooted maxillary anterior teeth and premolars that received 16 immediate implants equally randomized divided into 2 groups.
  control group: 8 implants were inserted in 8 fresh extraction sockets study group: 8 implants were inserted in 8 fresh extraction sockets followed by grafting with natural bovine bone substitute material with hyaluronic acid (act as study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): control group: 8 immediate implants were inserted in 8 fresh extraction sockets without bone grafting.
  Interventions: Combination Product: immediate dental implant
- study group (Active Comparator): study group: 8 immediate implants were inserted in 8 fresh extraction sockets followed by grafting with natural bovine bone substitute material with hyaluronic acid
  Interventions: Combination Product: immediate dental implant, natural bovine bone substitute material

INTERVENTIONS:
Combination Product: immediate dental implant — control group: 8 teeth were extracted then 8 immediate implants were placed without bone grafting
  Arms: control group
Combination Product: immediate dental implant, natural bovine bone substitute material — study group: 8 teeth were extracted then received 8 immediate implants followed by grafting with natural bovine bone substitute material with hyaluronic acid
  Arms: study group

SUMMARY:
the goal of this study is to evaluate the effective of natural bovine bone with hyaluronic acid on osseointegration of immediate implants in single rooted badly decayed maxillary anterior teeth and premolars. the main question it aims to answer is does natural bovine with hyaluronic acid affects osseointegration of immediate implants.

the study compares immediate implants followed by grafting with natural bovine bone with hyaluronic acid to immediate implants without grafting.

ELIGIBILITY:
Inclusion Criteria:

* medically free patients, good oral hygiene, no periapical lesions around teeth to be extracted

Exclusion Criteria:

* patients with bone or soft tissue defects, poor oral hygiene, heavy smoking, bruxism, severe periodontal disease

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Bone density | baseline (immediately) and 6 months
  using cone beam CT bone density was measured around the implant in housefield units immediately after implant placement and after 6 months.
implant stability | Baseline (immediately) and after 4 months
  using Osstell device, implant stability was measured immediately after implant placement and after 4 months

SECONDARY OUTCOMES:
Bone width | Baseline (immediately) and 6 months
  using cone beam CT, buccal bone width was measured from the mid surface of the implant immediately after implant placement and after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Said professor, Study Director — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: beginning when the data published with no end date